CLINICAL TRIAL: NCT00581321
Title: Acute Hemodynamic Effects of Oral Water in a Stable Cardiac Transplant Population
Brief Title: Oral Water Ingestion in Heart Transplant Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Satish R. Raj (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Satish R. Raj, Assistant Professor of Medicine & Cardiology, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 050811; UL1RR024975 (NIH)
Record Dates: First submitted 2007-12-22; First posted 2007-12-27 (Estimated); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Blood Pressure; Cardiac Transplantation
Keywords: water; blood pressure; vascular resistance; cardiac transplantation
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): water ingestion (16 fl oz within 3 minutes)
  Interventions: Dietary Supplement: water

INTERVENTIONS:
Dietary Supplement: water — water 500 ml x 1

SUMMARY:
In this study the investigators propose to assess the hemodynamic response to the ingestion of 16 fl oz of water. The investigators will test the hypothesis that water ingestion will increase the systemic vascular resistance.

DETAILED DESCRIPTION:
In this study we propose to assess the hemodynamic response to the ingestion of 16 fl oz of water. We will test the hypothesis that water ingestion will increase the systemic vascular resistance. This study will occur in patients status post cardiac transplantation during their clinical right heart catheterizations. Invasive hemodynamics including cardiac outputs and plasma norepinephrine levels will be measured before and 30 min after the water ingestion.

ELIGIBILITY:
Inclusion Criteria:

* s/p cardiac transplantation scheduled for clinical right heart catheterization
* age > 18 years

Exclusion Criteria:

* significant tricuspid regurgitation
* inability to safely swallow 500 ml of water
* other major medical comorbidities such as advanced renal disease where water ingestion may be harmful to patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-01; Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
change in total vascular resistance | 40 min (before to 30 min after water ingestion
  TPR measured by Modelflow

SECONDARY OUTCOMES:
blood pressure | 40 min
  peak BP over 40 min
heart rate | 40 min
  HR at time of peak BP over 40 min
plasma norepinephrine | 40 minutes
  plasma norepinephrine drawn 40 min post ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Tennessee Valley Health Systems (Nashville VA), Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee